CLINICAL TRIAL: NCT02540291
Title: An Open-Label Multicenter Phase 1 Study of E7046 in Subjects With Selected Advanced Malignancies
Brief Title: Study of E7046 in Subjects With Selected Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to, licensing agreement granting exclusive rights of research, development, manufacture and marketing of Eisai's E7046 to Adlai Nortye Biopharma.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7046-G000-101; 2014-004823-37 (EudraCT Number)
Record Dates: First submitted 2015-08-25; First posted 2015-09-03 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2018-07

CONDITIONS: Tumors
Keywords: E7046; Advanced malignancies; malignancies
MeSH Terms: conditions — Neoplasms | interventions — E7046

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E7046 (Experimental): Participants with tumor types that harbor high levels of myeloid infiltrate based on the Cancer Genome Atlas (TCGA).
  Interventions: Drug: E7046

INTERVENTIONS:
Drug: E7046 — E7046 will be administered as a single agent orally once daily (QD) continuously in 21-day cycles. In the dose escalation part, increasing doses of E7046 ranging from 125 mg to 750 mg will be administered to cohorts of 6 participants. In the cohort expansion part, participants will be treated at the RP2D.

SUMMARY:
This is an open label, multicenter, Phase 1 study of E7046 to assess the safety and tolerability of E7046 and to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of E7046.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts: a dose escalation part to determine the MTD and/or RP2D of E7046, and a cohort expansion part with 6 to 16 participants to better characterize safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) at the RP2D. In the dose escalation part, increasing doses of E7046 will be administered to cohorts of 6 participants, at dose levels ranging from 125 mg to 750 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
3. Life expectancy greater than or equal to 12 weeks
4. Participants must have any of the following tumor types, confirmed by available pathology records or current biopsy, that is advanced, nonresectable, or recurrent and progressing since last antitumor therapy, and for which no alternative standard therapy exists: pancreatic adenocarcinoma, renal clear cell carcinoma, SCCHN (squamous cell carcinoma of head and neck), NSCLC (non-small cell lung cancer), colorectal cancer (CRC), hepatocellular carcinoma (HCC), ovarian serous epithelial cancer, bladder transitional cancer, cervical cancer, and triple-negative breast cancer
5. Prior chemotherapy or immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) must have been completed at least 4 weeks before study drug administration, and all adverse events (AEs) have either returned to baseline or stabilized
6. Prior definitive radiation therapy must have been completed at least 6 weeks before study drug administration and the irradiated lesions should show evidence of progression if they are intended to be considered target lesions. Prior palliative radiotherapy must be completed at least 2 weeks before study drug administration. The radiotherapy-related side effects must have resolved before the study entry. No radiopharmaceuticals (strontium, samarium) will be allowed within 8 weeks before study drug administration.
7. Participants must have accessible tumors and consent to repeated biopsy for performance of correlative tissue studies
8. Must have at least one measurable lesion per irRECIST (immune-related Response Evaluation Criteria Criteria in Solid Tumors):

   * At least 1 lesion of greater than or equal to 10 mm in the longest diameter for a non-lymph node or greater than or equal to 15 mm in the short-axis diameter for a lymph node that is serially measurable according to irRECIST using computerized tomography/magnetic resonance imaging (CT/MRI)
   * Lesions that have had definitive external beam radiotherapy or locoregional therapies such as radiofrequency (RF) ablation or brachytherapy must show evidence of progressive disease to be deemed a target lesion
9. Prior treated brain or meningeal metastases must be without evidence of progression (confirmed by MRI) for at least 8 weeks and off immunosuppressive doses of systemic steroids (greater than 10 mg/day prednisone or equivalent) for at least 4 weeks before study drug administration
10. Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses greater than 7.5 to 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks before study drug administration.
11. Participants with prior Hepatitis B or C are eligible on the condition that participants have adequate liver function as defined by Inclusion Criterion number 16 and Exclusion Criterion number 5
12. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple gated acquisition (MUGA) scan
13. Adequate renal function defined as serum creatinine less than 1.5 X ULN (upper limit of normal) or use SI units or calculated creatinine clearance greater than or equal to 50 mL/min per the Cockcroft and Gault formula
14. Adequate bone marrow function:

    * Absolute neutrophil count (ANC) greater than or equal to 1500/mm3 (greater than or equal to 1.5 X 103/ul)
    * Platelets greater than or equal to 100,000/mm3 (greater than or equal to 100 X 109/L)
    * Hemoglobin greater than or equal to 9.0 g/dL
15. Adequate liver function:

    * Total bilirubin less than or equal to 1.5 X ULN except for unconjugated hyperbilirubinemia of Gilbert's syndrome
    * Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 X ULN (less than or equal to 5 X ULN if participant has liver metastases). If alkaline phosphatase is greater than 3 X ULN (in absence of liver metastases) or greater than 5 X ULN (in presence of liver metastases) AND the participant also is known to have bone metastases, the liver-specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of total alkaline phosphatase
16. Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) less than or equal to 1.5
17. Willing and able to comply with all aspects of the protocol
18. Provide written informed consent prior to any study-specific screening procedures
19. Females must not be lactating or pregnant at screening or baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug. All females will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrheic, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception, from the last menstrual period prior to initiation of treatment, during Treatment Cycles, and for 30 days after the final dose of study treatment, and have a male partner who uses a condom. Highly effective contraception includes:

    * Double barrier methods of contraception such as condom plus diaphragm or cervical/vault cap with spermicide
    * Placement of an intrauterine device
    * Established hormonal contraceptive methods: oral, injectable, or implant. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation. Female participants exempt from this requirement are participants who practice total abstinence or have a male partner who is vasectomized with confirmed azoospermia. If currently abstinent, the participant must agree to use a double barrier method as described above if they become sexually active during the Treatment Cycles, and for 30 days after study drug discontinuation
20. Male participants must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception and use a condom throughout the study period and for 90 days after study drug discontinuation)

Exclusion Criteria:

1. Other malignancy active within the previous 2 years except for basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast that has completed curative therapy
2. Participants with any active autoimmune disease (Appendix 2) or a documented history of autoimmune disease, poorly controlled asthma or history of syndrome that required systemic steroids or immunosuppressive medications, except for participants with vitiligo or resolved childhood asthma/atopy. Participants with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study.
3. Participants with inflammatory bowel disease
4. Known human immunodeficiency virus (HIV) infection
5. Active infection requiring therapy, including known positive tests for Hepatitis B surface antigen and hepatitis C virus (HCV) RNA
6. Major surgery within 4 weeks before the first dose of study drug
7. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids except inhaled or intranasal corticosteroids (with minimal systemic absorption)
8. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, or vomiting) that might impair the bioavailability of E7046
9. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the participant's participation in this study
10. Use of other investigational drugs within 28 days or at least 5 half-lives (whichever is shorter) before study drug administration
11. Prior exposure to drugs that are antagonists of colony stimulating factor-1 receptor (CSF1R) like but not limited to emactuzumab (RG7155) (Roche), PLX3397 (Plexicon), and JNJ40346627 (J & J)
12. Use of any live vaccines (eg, intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines) within 28 days
13. Prolongation of corrected QT [QTcF (Fridericia's corrected QT interval)] interval to greater than 480 msec when electrolytes balance is normal
14. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment (including oral anticoagulation)
15. Females who are pregnant (positive urine test) or breastfeeding
16. Any history of a medical condition or a concomitant medical condition that, in the opinion of the investigator, would compromise the subject's ability to safely complete the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Boston, Massachusetts
  - Houston, Texas
- Villejuif, Cedex, France

REFERENCES:
- [Derived] Hong DS, Parikh A, Shapiro GI, Varga A, Naing A, Meric-Bernstam F, Ataman O, Reyderman L, Binder TA, Ren M, Liu M, Dayal S, Siu AY, Sachdev P, Xu L, Bhagawati-Prasad V, Tchakov I, Ooi CE, Bao X, Marabelle A. First-in-human phase I study of immunomodulatory E7046, an antagonist of PGE2-receptor E-type 4 (EP4), in patients with advanced cancers. J Immunother Cancer. 2020 Jun;8(1):e000222. doi: 10.1136/jitc-2019-000222. PMID 32554609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 sites in the United States and 1 site in France from 30 July 2015 to 27 February 2018.
Pre-assignment Details: A total of 31 participants with advanced malignancies were enrolled, of which 30 participants received study treatment. The study was terminated before the start of the cohort expansion part. The discontinuation of participants from study is presented in the overall study table below.
Groups:
- E7046 125 mg: Participants received E7046 125 milligram (mg) capsules, orally, once daily, in continuous 21-day treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
- E7046 250 mg: Participants received E7046 250 mg capsules, orally, once daily, in continuous 21-day treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
- E7046 500 mg: Participants received E7046 500 mg capsules, orally, once daily, in continuous 21-day treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
- E7046 750 mg: Participants received E7046 750 mg capsules, orally, once daily, in continuous 21-day treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
Period: Overall Study
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
Started | 8 | 8 | 7 | 7
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 8 | 7 | 7
Not completed — Death | 7 | 7 | 5 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal Of Consent | 0 | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received at least 1 dose of study drug.
Groups:
- E7046 125 mg: Participants received E7046 125 mg capsules, orally, once daily, in continuous 21-day treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
- Total: Total of all reporting groups
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg | Total
Number analyzed (Participants) | 8 | 8 | 7 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.15) | 53.0 (17.10) | 54.4 (13.40) | 64.4 (10.18) | 55.5 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4 | 3 | 11
  Male | 8 | 4 | 3 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 7 | 7 | 7 | 7 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 6 | 7 | 5 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug (approximately up to 2 years)
Population: The FAS included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
Participants
  TEAEs | 8 | 7 | 6 | 7
  SAEs | 5 | 6 | 3 | 3

2. Primary Outcome: Maximum Tolerated Dose (MTD) of E7046
Time Frame: Cycle 1 (21 days)
Population: The dose limiting toxicity (DLT) evaluable set included all participants who were evaluable for the DLTs and had taken at least 1 dose of E7046.
Measure: Number; unit: mg
Groups:
- E7046: All Participants: Participants received E7046 125, 250, 500 or 750 mg capsules, orally, once daily, in continuous 21-day treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
Arm/Group | E7046: All Participants
Number analyzed (Participants) | 30
mg | NA — MTD could not be determined due to the absence of DLTs.

3. Primary Outcome: Recommended Phase 2 Dose (RP2D) of E7046
Description: Two RP2Ds were planned to be evaluated.
Time Frame: Cycle 1 (21 days)
Population: The DLT evaluable set included all participants who were evaluable for the DLTs and had taken at least 1 dose of E7046.
Measure: Number; unit: mg
Groups:
- E7046: All Participants: Participants received E7046 125 mg, 250 mg, 500 mg or 700 mg capsules, orally, once daily, in continuous 21-day treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
Arm/Group | E7046: All Participants
Number analyzed (Participants) | 30
mg
  RP2D 1 | 250
  RP2D 2 | 500

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the percentage of participants achieving a best overall response of confirmed immune-related partial response (irPR) + immune-related complete response (irCR), according to immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) v1.1, from first dose date until disease progression/recurrence.
Time Frame: From first dose date until disease progression/recurrence (approximately up to 2 years)
Population: The FAS included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from first dose date to the date of the first documentation of confirmed disease progression or death, whichever occurs first, according to irRECIST v1.1. PFS was calculated using Kaplan-Meier product-limit method and Greenwood Formula.
Time Frame: From first dose date to the date of the first documentation of confirmed disease progression or death (approximately up to 2 years)
Population: The FAS included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
months | 1.5 [1.1 to 4.0] | 1.4 [1.1 to 4.1] | 1.3 [1.2 to 1.6] | 1.3 [0.9 to NA] — Upper limit of confidence interval could not be calculated because of high number of participants that were censored from the analysis.

6. Secondary Outcome: Duration of Response (DOR)
Description: The DOR is defined as the time from the date of first documented confirmed irCR/irPR, according to irRECIST v1.1 until the first documentation of confirmed disease progression or death, whichever came first.
Time Frame: From the date of first documented confirmed irCR/irPR until the first documentation of confirmed disease progression or death (approximately up to 2 years)
Population: The FAS included all participants who received at least 1 dose of study drug. No participants had irCR or irPR; therefore, the DOR could not be determined.
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR is percentage of participants achieving best overall response of confirmed irCR, irPR, or immune-related stable disease (irSD) (lasting at least 5 weeks), according to irRECIST v1.1 from the first dose date until disease progression/recurrence.
Time Frame: From the first dose date until disease progression/recurrence (approximately up to 2 years)
Population: The FAS included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
percentage of participants | 25.0 [3.2 to 65.1] | 25.0 [3.2 to 65.1] | 0 [0 to 0] | 42.9 [9.9 to 81.6]

8. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The CBR is the percentage of participants achieving irPR + irCR + irSD (lasting at least 24 weeks), according to irRECIST v1.1 from first dose date until disease progression/recurrence.
Time Frame: From first dose date until disease progression/recurrence (approximately up to 2 years)
Population: The FAS included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (Baseline) up to 30 days after the last dose of study drug (approximately up to 2 years)
Arm/Group | E7046 125 mg | E7046 250 mg | E7046 500 mg | E7046 750 mg
All-Cause Mortality (participants affected / at risk) | 7/8 | 7/8 | 5/7 | 7/7
Serious Adverse Events (participants affected / at risk) | 5/8 | 6/8 | 3/7 | 3/7
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8 | 6/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E7046 125 mg (N=8) | E7046 250 mg (N=8) | E7046 500 mg (N=7) | E7046 750 mg (N=7)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E7046 125 mg (N=8) | E7046 250 mg (N=8) | E7046 500 mg (N=7) | E7046 750 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (5) | 3 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 3 (6) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (4) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT02540291/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT02540291/SAP_001.pdf